CLINICAL TRIAL: NCT02849145
Title: Study to Evaluation Interest of the Circulating Tumor DNA Dosage in Patient With Hepatic Metastatic Uveal Melanoma Candidate to Complete Resection (R0)
Brief Title: Evaluation Interest of the Circulating Tumor DNA Dosage in Patient With Hepatic Metastatic Uveal Melanoma Candidate to Complete Resection (ct DNA R0)
Acronym: ctDNA R0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2014-06
Record Dates: First submitted 2016-07-13; First posted 2016-07-29 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Uveal Melanoma
Keywords: Circulating tumor DNA
MeSH Terms: conditions — Uveal Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological/Vaccine (Experimental)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — 7,5 ml of patient peripherical blood will be collected at each blood sample.

SUMMARY:
Prospective, open labelled, monocentric trial to evaluation of the circulating tumor DNA rate in the blood, before and after curative resection of hepatic metastasis of uveal melanoma (HMUM) and during post-surgery follow-up

DETAILED DESCRIPTION:
The ct DNA R0 study is a prospective, open labelled, monocentric trial. The aim is to evaluate the circulating tumor DNA rate in the blood, before and after curative resection of hepatic metastasis of uveal melanoma (HMUM) and during post-surgery follow-up.

The patient will have a blood sample before and after the surgery and during the post-surgery follow-up. The patient will have a maximum of 10 blood samples during the 2 years of his follow-up of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old or more
2. Patient with hepatic injury of metastatic uveal melanoma eligible for curative surgery (R0).
3. No other distant metastasis (CT thoracic -abdomino -pelvic, bone scan).Measurable metastatic disease (echography, CT and/or MRI, FDG-PET, (fluoro- D-glucose integrated with computed tomography)).
4. Patient able to stand a blood collection.
5. Patient explanation given and consent information signed or by legal representative.

   Exclusion Criteria:
6. Patient without social protection / insurance..
7. Patient with hepatic metastasis unresectable by surgery
8. Patient with extra-hepatic metastasis.
9. Person deprived of liberty or under guardianship
10. Inability to submit to medical monitoring of the trial for reasons of geography, social or psychological.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Correlation between the circulating tumor DNA rate before/after surgery and the rate of effective complete resection | Up to one month
  Comparison the circulating tumor DNA rate before/after surgery and the rate of effective complete resection.

SECONDARY OUTCOMES:
stability of the circulating tumor DNA on 2 pre-surgery samples | Up to one month
  Comparison the circulating tumor DNA rate before/after surgery
Study of the correlation between the variation rate of the circulating tumor DNA at different points (T0, T1, T2, T3, T4 and Tn) and the apparition time of metastasis on hepatic MRI during the study follow-up. | two years
  Timepoints :
  T0 and T1 : before surgery T2 : 2 days after surgery T3 : 8 days after surgery T4 to T9 : every 4 months up to two years.
Detection of GNA11 or GNAQ mutation on one of the hepatic metastasis | Up to one month
  Search of GNA 11 or GNAQ mutation by Next Generation Sequencing techniques
Comparative study of the mutation profile of the ocular tumor if available, resected hepatic metastasis. | Up to one month
Histological study of the resected hepatic metastasis (inflammation, Ki 67, necrosis, fibrosis and vascularization, genomic analysis of the metastasis) | Up to one month
Detection of genetic factors for uveal melanoma | Up to one month
  Search of genetic factors for uveal melanoma to be used as predictive evidence of the clinical response for possible future treatment
Study of overall survival after HMUM resection | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Mariani, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Mariani P, Bidard FC, Rampanou A, Houy A, Servois V, Ramtohul T, Pierron G, Chevrier M, Renouf B, Lantz O, Gardrat S, Vincent-Salomon A, Roman-Roman S, Rodrigues M, Piperno-Neumann S, Cassoux N, Stern MH, Renault S. Circulating Tumor DNA as a Prognostic Factor in Patients With Resectable Hepatic Metastases of Uveal Melanoma. Ann Surg. 2023 Oct 1;278(4):e827-e834. doi: 10.1097/SLA.0000000000005822. Epub 2023 Feb 27. PMID 36847256